CLINICAL TRIAL: NCT04235660
Title: Yttrium-90 Radiation Segmentectomy Versus Stereotactic Body Radiation Therapy (SBRT) for the Treatment of Early Stage Hepatocellular Carcinoma (HCC): A Pilot Study
Brief Title: Y90 Radiation Segmentectomy vs SBRT for HCC
Acronym: SBRT vs Y90
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: unable to recruit. terminated due to futility
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Paul Haste, Assistant Professor of Clinical Radiology & Imaging Sciences, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IU-2001712954
Record Dates: First submitted 2020-01-15; First posted 2020-01-22 (Actual); Results first posted 2023-10-25 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Hepatocellular Carcinoma (HCC)
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiosurgery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Radiologist assessing response will be blinded to the treatment type
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Yttrium-90 Radiation Segmentectomy (Active Comparator)
  Interventions: Radiation: Yttrium-90 Radiation Segmentectomy
- Stereotactic Body Radiation Therapy (Active Comparator)
  Interventions: Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Radiation: Yttrium-90 Radiation Segmentectomy — This therapy arm involves two separate steps, a planning/mapping arteriogram and a therapy delivery. The planning arteriogram will be performed to confirm arterial anatomy is acceptable for RS (≤2 segment delivery) and that lung shunting is not too high to preclude treatment with RS. Once confirmed, patients will return for RS (within 45 days of mapping). Dose will be calculated based off the desired treatment volume using pre-treatment cross-sectional imaging. The desired segmental dose will be calculated to be ≥ 200Gy. RS will be performed by one of three separate interventional radiologists with experience in radioembolization. Actual administered activity and location of dose administration will be recorded.
  Arms: Yttrium-90 Radiation Segmentectomy
Radiation: Stereotactic Body Radiation Therapy — SBRT will be delivered with linear accelerator-based photon beams with either fixed angle non- coplanar fields or dynamic arcs. An internal target volume (ITV) will be generated to account for tumor movement during breathing cycle. Finally, a planning target volume (PTV) will be an expansion of 3- 5mm from the ITV. For Child Pugh A patients, prescription dose will either be 5000cGy in 5 fractions delivered every other day or 4800cGy in 3 fractions delivered twice weekly. For Child Pugh B patients, prescription dose of 4000cGy in 5 fractions delivered every other day. Inverse planning will be used. 95% of the PTV or more will receive at least 100% of the prescription dose. Normal tissue dose constraints for each dose level will be respected with acceptable deviations permitted as outlined in appendix VII. Patients will be seen at least once per week by a clinician to grade toxicities, with on- treatment labs (CBC, CMP, INR) each week.
  Arms: Stereotactic Body Radiation Therapy

SUMMARY:
The proposed study is a single site, prospective, randomized pilot study to assess the feasibility of recruitment of patients into a trial evaluating the efficacy and tolerability of selective transarterial Y90 radioembolization (radiation segmentectomy) versus stereotactic body radiation therapy (SBRT) for solitary early stage (≤ 3cm) hepatocellular carcinoma (HCC).

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and HIPAA authorization
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male or female, aged ≥ 18 years at time of informed consent
* Solitary HCC (≤3 cm) diagnosed by imaging (LI-RADS 4-5) or histology
* Childs-Pugh score ≤ 7
* ECOG performance status 0-1
* Tumor location/characteristics eligible for either SBRT or Y90 therapy as deemed by local tumor board
* Adequate organ function defined as:

  1. serum bilirubin < 4.0 mg/dL ,
  2. albumin > 2 g/dL

Exclusion Criteria:

* Any prior locoregional therapy to the target tumor
* Any prior radiation therapy to the liver
* Pregnancy or lactation: Women of childbearing potential must have a negative pregnancy test within 14 days of protocol registration. Women are considered to have childbearing potential (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) unless they meet one of the following criteria:

  i. Has undergone a hysterectomy or bilateral oophorectomy; or ii. Has been naturally amenorrheic for at least 24 consecutive months
* Known severe allergic reaction (anaphylaxis) to iodinated contrast
* Coagulopathy (platelets < 50 K/mm3 and/or INR > 2) not correctable by transfusion
* Macrovascular invasion or extrahepatic HCC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-07-22 (Actual); Primary Completion 2022-03-08 (Actual); Study Completion 2022-03-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Yttrium-90 Radiation Segmentectomy | Stereotactic Body Radiation Therapy
Started | 1 | 1
Completed | 0 | 0
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Yttrium-90 Radiation Segmentectomy | Stereotactic Body Radiation Therapy | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Recruitment (Recruitment Rate)
Description: Feasibility of recruitment will be measured by evaluating the proportion of patients enrolled versus those approached for the study after they have been determined to be a candidate.
Time Frame: 24 months
Population: This group consists of all patients who fit inclusion/exclusion criteria and were approached for enrollment in the study
Measure: Count of Participants; unit: Participants
Groups:
- Eligible Participants: This group consists of all patients who fit inclusion/exclusion criteria and were approached for enrollment in the study
Arm/Group | Eligible Participants
Number analyzed (Participants) | 22
Participants
  recruited | 2
  declined to participate | 20

2. Secondary Outcome: Proportion of Patients With Any Toxicities
Description: the proportion of patients with any toxicities (≥ grade 4) using CTCAE between RS and SBRT for patients with small (≤3 cm) solitary hepatocellular carcinoma (HCC).
Time Frame: 16 months for the first subject and 4 months for the second
Population: No data were collected for this outcome measure because 0 participants remained enrolled in this time frame
Arm/Group | Yttrium-90 Radiation Segmentectomy | Stereotactic Body Radiation Therapy
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Mean Change in Hepatobiliary Function
Description: the mean change in hepatobiliary function, as measured 3 months after treatment using a functional HIDA scan, between RS and SBRT for patients with small (≤3 cm) solitary hepatocellular carcinoma (HCC).
Time Frame: 16 months for the first subject and 4 months for the second
Population: 1 pt in y90 arm had 3 month scan to compare to baseline. no other scans
Measure: Number; unit: percentage of liver function decrease
Arm/Group | Yttrium-90 Radiation Segmentectomy | Stereotactic Body Radiation Therapy
Number analyzed (Participants) | 1 | 0
percentage of liver function decrease | 9.1 |

4. Secondary Outcome: Mean Change in Functional Assessment of Cancer Therapy- General (FACT-G) Score
Description: the mean change in patient-reported outcomes from baseline, at 1, 3 and 6 months, between RS and SBRT, for patients with small (≤3 cm) solitary hepatocellular carcinoma (HCC), using the Functional Assessment of Cancer Therapy- General (FACT-G). scale goes from 0-108 with a higher score being better.
Time Frame: 6 months
Population: for single Y90 pt data was collected. Data not collected for SBRT pt.
Measure: Number; unit: score on a scale
Arm/Group | Yttrium-90 Radiation Segmentectomy | Stereotactic Body Radiation Therapy
Number analyzed (Participants) | 1 | 0
score on a scale
  base line score | 69 |
  1 month | 75 |
  3 month | 82 |
  6 month | 78 |

5. Secondary Outcome: Mean Change in Comprehensive Score for Financial Toxicity
Description: the mean change in patient-reported outcomes from baseline, at 1, 3 and 6 months, between RS and SBRT, for patients with small (≤3 cm) solitary hepatocellular carcinoma (HCC), using the Comprehensive Score for Financial Toxicity (COST). scale is from 0-44 with higher being bettter
Time Frame: 6 months
Population: data collected for single y90 pt. data not collected for SBRT pt
Measure: Number; unit: score on a scale
Arm/Group | Yttrium-90 Radiation Segmentectomy | Stereotactic Body Radiation Therapy
Number analyzed (Participants) | 1 | 0
score on a scale
  baseline | 27 |
  1 month | 29 |
  3 month | 23 |
  6 month | 16 |

6. Secondary Outcome: Disease-free Survival (DFS) Rates of RS and SBRT
Description: the disease-free survival (DFS) rates of RS and SBRT at 2 years using mRECIST on CT or MR for patients with small (≤3 cm) solitary hepatocellular carcinoma (HCC).
Time Frame: 16 months for the first subject and 4 months for the second
Population: No data were collected for this outcome measure because 0 participants remained enrolled in this time frame
Arm/Group | Yttrium-90 Radiation Segmentectomy | Stereotactic Body Radiation Therapy
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Time-to-secondary Treatment (TTST) Between RS and SBRT
Description: time-to-secondary treatment (TTST) between RS and SBRT for patients with small (≤3 cm) solitary hepatocellular carcinoma (HCC) up to 2 years after initial treatment.
Time Frame: 16 months for the first subject and 4 months for the second
Population: No data were collected for this outcome measure because 0 participants remained enrolled in this time frame
Arm/Group | Yttrium-90 Radiation Segmentectomy | Stereotactic Body Radiation Therapy
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Objective Response Rate
Description: the objective response rate (ORR) of radiation segmentectomy (RS) and stereotactic body radiation therapy (SBRT) as measured at 6 months using mRECIST (appendix IV) for patients with small (≤3 cm) solitary hepatocellular carcinoma (HCC) to better allow for an appropriately powered trial evaluating the efficacy of these treatments.
Time Frame: 6 months
Population: No data were collected for this outcome measure because 0 participants in the SBRT arm remained enrolled in this time frame and 6 month imaging was unavailable for the pt in the y90 arm
Arm/Group | Yttrium-90 Radiation Segmentectomy | Stereotactic Body Radiation Therapy
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: adverse event data was planned to be collected for up to 24 months. however, total AE data only collected for 15 months from enrollment (at the longest) secondary to pt drop out.
Arm/Group | Yttrium-90 Radiation Segmentectomy | Stereotactic Body Radiation Therapy
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Yttrium-90 Radiation Segmentectomy (N=1) | Stereotactic Body Radiation Therapy (N=1)
fatigue (General disorders) | 1 | 1 — grade 1 fatigue
nausea (Gastrointestinal disorders) | 1 | 0 — grade 1
right leg bruise (Surgical and medical procedures) | 1 | 0 — grade 1 bruise
elevated vitamin D (General disorders) | 1 | 0 — grade 1
elevated AFP (Hepatobiliary disorders) | 1 | 0 — grade 1
elevated AST (Hepatobiliary disorders) | 1 | 0 — grade 1
low serum carbon dioxide (General disorders) | 1 | 0 — grade 1
high anion gap (General disorders) | 1 | 0 — grade 1
decreased lymphocyte count (Blood and lymphatic system disorders) | 1 | 0 — grade 1
decreased platelet count decreased (Blood and lymphatic system disorders) | 1 | 0 — grade 1
glucose intolerance (General disorders) | 1 | 0 — grade 1
ALT increased (General disorders) | 1 | 0 — grade 1
perirectal abscess (General disorders) | 1 | 0 — grade 2
increased size of left renal mass (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 — grade 1
low sodium (General disorders) | 1 | 0 — grade 1
decreased lymphocyte count (Blood and lymphatic system disorders) | 1 | 0 — grade 2
decreased lymphocyte count (Blood and lymphatic system disorders) | 1 | 0 — grade 3
abdominal pain (Gastrointestinal disorders) | 0 | 1 — grade 2
low creatinine (General disorders) | 0 | 1 — grade 1

LIMITATIONS AND CAVEATS:
This study was originally planned as a pilot in hopes of being able to demonstrate feasibility of recruitment into a trail where one arm involved invasive therapy and one non-invasive. Unfortunately, the trial opened very shortly after the beginning of the pandemic in 2020 and overall recruitment/resources for research were hindered. after close to 18 months with little enrollment the funding entity and research team agreed it should just be terminated early for futility.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-15): https://cdn.clinicaltrials.gov/large-docs/60/NCT04235660/Prot_SAP_001.pdf